CLINICAL TRIAL: NCT06556667
Title: Comparison of Maximum Energy Shocks From Two Defibrillator Vendors MAX - SHOCK- A Randomized Controlled Clinical Trial
Brief Title: MAX - SHOCK Clinical Trial
Acronym: MAX-SHOCK
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ottawa Heart Institute Research Corporation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: CRRF 6004
Record Dates: First submitted 2024-07-31; First posted 2024-08-16 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Cardioversion; Atrial Fibrillation
Keywords: defibrillator
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Intervention Model Description: two arms will be compared using the Chi squared test
Who Masked: Participant
Masking Description: participants will not know which defibrillator was used during their cardioversion.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 200J (Active Comparator): biphasic defibrillator with maximum energy of 200J (® Zoll)
  Interventions: Device: biphasic defibrillator with maximum energy of 200J (® Zoll)
- 360J (Active Comparator): biphasic defibrillator with maximum energy of 360J (® Physio-Control)
  Interventions: Device: biphasic defibrillator with maximum energy of 360J (® Physio-Control)

INTERVENTIONS:
Device: biphasic defibrillator with maximum energy of 200J (® Zoll) — Cardioversion
  Arms: 200J
Device: biphasic defibrillator with maximum energy of 360J (® Physio-Control) — Cardioversion
  Arms: 360J

SUMMARY:
Can Electrical Cardioversion (ECV) for AF be improved. It is the preferred method to restore sinus rhythm in patients with AF in whom a rhythm-control strategy is pursued.

Hypothesis:

ECV success rates will be greater with a biphasic defibrillator with maximum energy of 360J (® Physio-Control) compared to a biphasic defibrillator with maximum energy of 200J (® Zoll)

DETAILED DESCRIPTION:
Published estimates of ECV success using modern biphasic defibrillators vary considerably but most are limited by small sample sizes. Our pre-intervention ECV success rate of 91.8% was stable over >2.5 years and is comparable to a previous study from our institute11 and to recent estimates from moderately sized studies using contemporary technology. For instance, the Euro Heart Survey on AF reported an ECV success rate of 91% in 424 patients2 and the Biphasic Energy Selection for Transthoracic cardioversion of Atrial Fibrillation (BEST AF) trial reported 89% success in 380 patients.3 The variability in starting shock energy and shock energy escalation observed at our centre prior to implementing the OAFCP is also consistent with reported practices elsewhere. A recent survey of 57 European centres found that nearly two-thirds of hospitals started with a 100 J biphasic shock for AF whereas the remaining third started with 200 J.1 Considerable differences in electrode placement were also reported in this survey with 58.7% of centres using an anterolateral position and the remainder using an anteroposterior approach.1Our investigators and others have previously shown that physicians seldom apply sufficient force even when prompted to do so and even when using handheld paddles.10,16,17 ECV practices at our institute prior to implementing the OAFCP were therefore likely representative of those at most centres.

ELIGIBILITY:
Inclusion Criteria:

* Patients age > 18 years.
* Persistent atrial fibrillation.
* Scheduled for elective cardioversion at UOHI
* Patient is within the circle of care of UOHI Electrophysiology staff

Exclusion Criteria:

* Known left-atrial appendage thrombus.
* Contraindication to appropriate anticoagulation.
* Patient is included in another randomized clinical trial.
* Patient does not meet all of the above listed inclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 376 (Estimated)
Dates: Start 2025-03-31 (Actual); Primary Completion 2027-09-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
ECV success | 2 seconds
  ECV success defined as >_2 consecutive sinus beats, or captured atrial-paced beats in patients with implanted cardiac devices, after shock delivery

SECONDARY OUTCOMES:
First shock success | 2 seconds
  Cardioversion is successful without crossover
sustained success | 4 hours
  sustained sinus or atrial paced rhythm documented on 12-lead electrocardiogram

CONTACTS AND LOCATIONS:
Overall Officials: Mehrdad Golian, Principal Investigator — Ottawa Heart Institute Research Corporation
Locations (1):
- University of Ottawa Heart Institute, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No